CLINICAL TRIAL: NCT04877288
Title: A Prospective, Open-label, Multicenter, Randomized Study to Evaluate the Benefits and Risks of Conversion of Existing Adolescent Renal Allograft Recipients Aged 12 to Less Than 18 Years of Age to a Belatacept-based Immunosuppressive Regimen as Compared to Continuation of a Calcineurin Inhibitor-based Regimen, and Their Adherence to Immunosuppressive Medications
Brief Title: A Study to Evaluate the Benefits and Risks of Conversion of Existing Adolescent Kidney Transplant Recipients Aged 12 to <18 Years to a Belatacept-based Immunosuppressive Regimen as Compared to Continuation of a Calcineurin Inhibitor-based Regimen, and Their Adherence to Immunosuppressive Medications
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IM103-402; 2022-501677-39 (Other: EU CTR)
Record Dates: First submitted 2021-05-03; First posted 2021-05-07 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Renal Allograft Recipients
Keywords: Acute rejection; Belatacept; Calcineurin inhibitors (cyclosporine, tacrolimus); Conversion; Donor-specific antibodies; eGFR; Immunosuppressive regimen; Adolescent kidney transplant recipients
MeSH Terms: interventions — Abatacept; Tacrolimus; Cyclosporine; Mycophenolic Acid; Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1: Conversion from a CNI- to belatacept-based regimen after a period of overlap (Experimental): Conversion followed by tapering and discontinuation of the calcineurin inhibitor (CNI)
  Interventions: Biological: Belatacept; Drug: Tacrolimus; Drug: Cyclosporine A; Drug: Mycophenolate Mofetil; Drug: Enteric Coated Mycophenolate Sodium; Drug: Corticosteroids
- Arm 2: Continue calcineurin inhibitor-based regimen (Active Comparator)
  Interventions: Drug: Tacrolimus; Drug: Cyclosporine A; Drug: Mycophenolate Mofetil; Drug: Enteric Coated Mycophenolate Sodium; Drug: Corticosteroids

INTERVENTIONS:
Biological: Belatacept — Specified dose on specified days
  Other Names: Nulojix
  Arms: Arm 1: Conversion from a CNI- to belatacept-based regimen after a period of overlap
Drug: Tacrolimus — Specified dose on specified days
Drug: Cyclosporine A — Specified dose on specified days
Drug: Mycophenolate Mofetil — Specified dose on specified days
Drug: Enteric Coated Mycophenolate Sodium — Specified dose on specified days
Drug: Corticosteroids — Specified dose on Specified days

SUMMARY:
The purpose of this study is to evaluate the benefits and risks of conversion of existing adolescent kidney allograft recipients aged 12 to less than 18 years of age to a belatacept-based immunosuppressive regimen as compared to continuation of a calcineurin inhibitor-based regimen and their adherence to immunosuppressive medications.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adolescents 12 to less than 18 years of age
* Recipients of a renal allograft from a living or deceased donor transplanted at least 6 calendar months prior to enrollment
* Receiving a stable regimen of a calcineurin inhibitor (CNI), with mycophenolate mofetil (MMF) or enteric-coated mycophenolate sodium/mycophenolate mofetil (EC-MPS/MPA), with or without daily corticosteroids for ≥ 30 days prior to randomization
* Clinically stable renal function during the 12-week period prior to screening, in the opinion of the investigator and based on protocol-defined criteria for proteinuria and estimated glomerular filtration rate (eGFR)
* Serologic evidence of past exposure to Epstein-Barr virus (EBV) and current absence of EBV DNA replication at or prior to renal transplantation and during the Screening period
* Completion of an initial course of SARS-CoV-2 vaccination per local standard of care, a minimum of 6 weeks prior to enrollment

Exclusion Criteria:

* Recipients with EBV serostatus negative or unknown at screening or at transplant
* Treatment for biopsy-proven acute rejection (BPAR) of any degree of severity within 6 calendar months prior to enrollment
* Biopsy-confirmed antibody-mediated acute rejection at any time with the current allograft
* Banff 97 grade IIA or higher acute cellular rejection (or equivalent), or treatment with plasmapheresis or rituximab for any acute rejection at any time with the current allograft
* Current evidence or past history of active or inadequately treated latent tuberculosis (TB) infection
* Previously treated with belatacept or previously enrolled in a belatacept trial with their present allograft

Other inclusion/exclusion criteria apply

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 102 (Estimated)
Dates: Start 2021-07-21 (Actual); Primary Completion 2032-12-30 (Estimated); Study Completion 2034-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants who survive with a functional graft with estimated glomerular filtration rate (eGFR) > 30 mL/min/1.73 m2 (updated Schwartz formula) at 24 months post-randomization | 24 months

SECONDARY OUTCOMES:
Participant and graft survival: Proportion of participants who survive with a functioning graft | 6, 12 and 24 months
Participant and graft survival: Proportion of participants who survive | 6, 12, and 24 months
Participant and graft survival: Proportion of participants who experience death-censored graft loss | 6, 12, and 24 months
Acute rejection: Incidence of clinically suspected biopsy-proven acute rejection (BPAR) | 3, 6, 12, and 24 months
Acute rejection: Severity of clinically suspected, biopsy confirmed rejection as determined by locally and centrally reviewed histopathology | 3, 6, 12, and 24 months
Renal function as assessed by: Serum creatinine concentration | Up to 24 months
Renal function as assessed by: Estimated GFR (eGFR per updated Schwartz combined equation) | Up to 24 months
Renal function as assessed by: eGFR per updated bedside Schwartz approximating equation | Up to 24 months
Renal function as assessed by: eGFR per Full Age Spectrum (FAS) equation of Potell et al | Up to 24 months
Renal function as assessed by: eGFR per age and sex-dependent equation of Pierce et al | Up to 24 Months
Proteinuria, as assessed by urinary protein:creatinine ratio (UPCR), as determined from single-voided urine specimens | Up to 24 months
Slope of change in eGFR over time, as assessed by baseline-adjusted mean eGFR determinations at protocol-specified study visits | Up to 24 months
Adherence to immunosuppressive medications as assessed by variation in calcineurin inhibitor pre-dose whole blood concentrations by summaries over time of monitored adherence to orally administered immunosuppressive medications | up to 24 months
Adherence to immunosuppressive medications, as assessed by: Variations in pre-dose concentrations of calcineurin inhibitor in whole blood | Up to 24 months
Adherence to immunosuppressive medications, as assessed by: 7-day recall of missed and late doses of each orally administered immuno-suppressive medication at protocol-specified study visits | Up to 24 months
Adherence to immunosuppressive medications, as assessed by: Monitoring of compliance with monthly belatacept infusions | Up to 24 months
Adherence to immunosuppressive medications, as assessed by: Periodic review of parents' and patients' perceived barriers to adherence to the prescribed immunosuppressive medications regimen | Up to 24 months
Mean blood pressure over time | Up to 24 months
Mean blood pressure changes from baseline over time | Up to 24 months
Intensity of antihypertensive drug therapy, defined as the total number of medications used to maintain BP control | Up to 24 months
Monitoring of safety laboratory parameters over time: Mean fasting lipid profiles | Up to 24 months
Monitoring of safety laboratory parameters over time: Fasting blood glucose concentrations | Up to 24 months
Monitoring of safety laboratory parameters over time: Hemoglobin A1c concentrations | Up to 24 months
Donor Specific antibodies (DSA): Proportion of participants with pre-existing anti-human leukocyte antigen (HLA) DSAs at baseline and with de novo anti-HLA DSA post-randomization | 6, 12, and 24 months
Immunogenicity of belatacept as determined by the proportion of participants with detectable serum anti-belatacept antibodies | 6, 12, and 24 months
Belatacept pre-dose (C0) serum concentrations | Up to 24 months
Mean percent belatacept CD86 receptor occupancy | Baseline
Post-randomization changes from baseline percent belatacept CD86 receptor occupancy | 6, 12, and 24 months
Safety and tolerability of belatacept following conversion: Incidence of Adverse Events (AEs) | up to 24 months
Safety and tolerability of belatacept following conversion: Incidence of Serious Adverse Events (SAEs) | Up to 24 months
Safety and tolerability of belatacept following conversion: Incidence of laboratory marked abnormalities | Up to 24 months
Proportion of participants within each stage of the Tanner staging scale | Up to 24 months
  The Tanner scale is a measure of pubertal development (sexual maturation) in children and adolescents with components described for each sex, rated separately on a scale of stage one to stage five, with 1 for preadolescent and 5 for mature/adult
Linear growth (height) | Up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (38):
- United States (15):
  - Local Institution - 0042, Birmingham, Alabama
  - Local Institution - 0041, Los Angeles, California
  - Local Institution - 0014, Washington D.C., District of Columbia
  - Local Institution - 0022, Hollywood, Florida
  - Local Institution - 0045, Miami, Florida
  - Local Institution - 0049, Atlanta, Georgia
  - Local Institution - 0033, Chicago, Illinois
  - Local Institution - 0017, Baltimore, Maryland
  - Local Institution - 0044, Boston, Massachusetts
  - Local Institution - 0043, St Louis, Missouri
  - Local Institution - 0024, Durham, North Carolina
  - Local Institution - 0025, Cincinnati, Ohio
  - Local Institution - 0048, Cleveland, Ohio
  - Local Institution - 0052, Portland, Oregon
  - Local Institution - 0038, Seattle, Washington
- Argentina (2):
  - Local Institution - 0060, ABB, Buenos Aires F.D.
  - Local Institution - 0062, Buenos Aires
- UZ Gent-Paediatric Nephrology and Rheumatology Department, Ghent, Belgium
- France (6):
  - Centre Hospitalier Universitaire de Nantes - L' Hopital l'hôtel-Dieu, Nantes, Loire-Atlantique
  - Bordeaux University Hospital - Pellegrin-Pediatrics, Bordeaux
  - Hospices Civils de Lyon - Hôpital Femme Mère Enfant-néphrologie pédiatrique, Bron
  - Hopital De La Timone, Marseille
  - Hopital Necker, Paris
  - Assistance Publique - Hopitaux de Paris (AP-HP) - Hopital Robert Debre - Centre Hospitalo Universita, Paris
- Germany (4):
  - Universitaetsklinikum Essen, Essen, North Rhine-Westphalia
  - Universitaetsklinikum Koeln-Klinik und Poliklinik für Kinder- und Jugendmedizin, Abteilung für Pädia, Cologne
  - Local Institution - 0011, Hamburg
  - Local Institution - 0026, Heidelberg
- Italy (3):
  - IRCCS Istituto Giannina Gaslini, Genoa, Liguria
  - Local Institution - 0030, Milan
  - Ospedale Regina Margherita-S.C Nefrologia, Dialisi e Trapianto Renale, Torino
- Emma Children (AMC), Amsterdam, Netherlands
- Local Institution - 0061, Oslo, Norway
- Spain (3):
  - Local Institution - 0001, Barcelona
  - Local Institution - 0012, Rivas-Vaciamadrid
  - Local Institution - 0003, Seville
- United Kingdom (2):
  - Local Institution - 0008, Manchester
  - Queen's Medical Centre, Nottingham University Hospitals-Children's Clinical Research Team, Nottingham

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT04877288.html